CLINICAL TRIAL: NCT03620968
Title: "Implementation of a Cognitive Training Program in the Elderly to Reduce the Risk of Postoperative Cognitive Dysfunction in Elective Non-cardiac Surgery "
Brief Title: Implementation of a Cognitive Training Program to Reduce the Risk of Postoperative Cognitive Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Medico Teknon (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Bibiana Ros Nebot, MSN, RN Anesthesia Nurse, Centro Medico Teknon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DCPO2017
Record Dates: First submitted 2017-12-26; First posted 2018-08-08 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Postoperative cognitive dysfunction; Cognitive training; Anaesthesia in Non-cardiac surgery; Elderly adult; Perioperative management.
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (No Intervention): Control, no intervention
- Group 2 (Experimental): Intervention before surgery (cognitive training)
  Interventions: Other: cognitive training
- Group 3 (Experimental): Intervention Before and after surgery (cognitive training)
  Interventions: Other: cognitive training

INTERVENTIONS:
Other: cognitive training — 15 minutes day of brain training by an APP
  Arms: Group 2; Group 3

SUMMARY:
Background: The postoperative cognitive dysfunction (POCD) is a frequent complication, often underestimated and leads to a negative impact on the quality of life for patients and their families.

Objective: Measure the effectiveness of the cognitive training in reducing POCD in patients 55 and 70 years old undergoing elective non cardiac surgery with a degree II-III (medium-high) in "Centro Médico Teknon" Barcelona, during 2017-2018.

Methodology: Randomized control clinical trial. The anticipate sample size is approximately 225, 75 in each group. Cognitive training performed at different stages of the perioperative period. Measure the cognitive function through a battery of neuropsychological tests during the preoperative (10 days pre-surgery) and postoperative (at 3 - 30 and 90 days post-surgery). Data analysis: SPSS 22, descriptive and inferential analysis: Chi-square, Student's t-test, ANOVA and Pearson correlation (p<0,05).

Limitations: Loss for non-intervention and loss of follow-up. Applicability: Strategy to improve the quality of life patients and reduce socioeconomic costs associated.

DETAILED DESCRIPTION:
Postoperative Cognitive Dysfunction (PCD) is a frequent and serious complication associated with the surgical / anesthetic act. It is an under-recognized and underestimated entity, as it can often go unnoticed even though its effects can be devastating. The cognitive domains affected are diverse and can include memory, perception, verbal abilities and executive functions.

It is not the only postoperative cognitive disorder and for this reason it is important not to confuse it with delirium and dementia. Cognitive dysfunction still does not have a diagnostic code formally defined by ICD-10 (International Classification of Disease) or by the DSM-V, although the medical field has begun to use this term for the general description of those patients who complain about memory alterations and the thought process in the postoperative period. Its detection and evaluation depend on the comparative analysis of the cognitive function (analyzed by means of neuropsychological tests) betinestigatorsen the pre and postoperative period. It is considered, in most of the cases, a mild or moderate cognitive impairment of a transient and reversible nature. Its etiology is unknown, and it is related to a complex and multifactorial pathophysiology. The most accepted physiopathological hypothesis is the inflammatory alteration of the Central nervous system (neuroinflammation) due to surgical trauma, with the consequent deterioration of the cognitive reserve contributing to a cognitive deficit. At the present moment there is no effective strategy tested to prevent PCD.

Some of the most relevant studies on this disorder inestigatorsre published in The Lancet in 1998 (Moller et al.) and Anesthesiology in 2008 (Monk et al.). These studies determined that surgery and anesthesia caused PCD in the long term. They also concluded that the PCD appears in all ages but that old age exponentially increases the risk of suffering it. In addition, a low educational level increases the risk of PCD and people who maintain a PCD after 3 months, are more likely to experience dementia and a higher mortality risk in the first year after surgery.

The relevant impact of this disorder is dependent on an increase in mortality, a workforce loss due to incapacity and early retirement, and social cost due to sick leave, medical and nursing homes for the, now dependent, patient.

At present, it is important to identify, create and evaluate procedures aimed at helping patients at risk from this disorder from anesthesia consultations, as a way to help improve the outcomes. In this sense, this project proposes the validation of cognitive training as a non-pharmacological intervention to reduce incidence and intensity of Postoperative Cognitive Dysfunction.

This intervention is based on the fact that an increase in the neurological functional reserve could serve as a protective factor against cognitive dysfunction, improving plasticity and brain reserve and subsequently improving the performance of mental capacities, through organized techniques and exercises before surgery. It is proposed as the first non-pharmacological intervention in cases of normal aging, mild cognitive impairment and slight dementia. In addition, it´s low cost and has no significant negative effects.

Therefore, inestigators propose a cognitive training APP, developed by Spanish Neuropsychologists aimed at improving cognitive functions, that can be accessed from an online platform meant for practitioners to oversee patient development.

Main objective: Measure the effectiveness and impact of the cognitive training program "Sincrolab" on Postoperative Cognitive Dysfunction in patients aged 55-70 years, after elective, non-cardiac, degree-II-III complexity (mid-high), surgery, in Centro Médico Teknon, Barcelona, betinestigatorsen 2019-2020

Specific objectives:

1. Measure the incidence of PCD in different study groups at 3 days, 1 month and 3 months of the surgical procedure.
2. Compare the evolution of PCD in the intervention group and the control group.
3. Measure the duration and intensity of the PCD in the different study groups.
4. Identify the development of PCD in relation to: age, sex, the type of surgical intervention, duration of surgery, types of anesthesia, postoperative complication.
5. Measure the adherence to the proposed cognitive training pattern, determining the rate of drop-outs.

Study Hypothesis The implementation of a cognitive training program during the perioperative period decreases the incidence, intensity and duration of Postoperative Cognitive Dysfunction.

Design of the study:

It is an epidemiological study, located in the empirical-analytic paradigm, that intends to obtain knowledge objectively identifying, the cause-effect relationships betinestigatorsen cognitive training during the perioperative and the development of PCD, by studying memory alterations and executive functions. It's a pre-test/post-test experimental study design, with random allocation, and the creation of 3 study groups:

1. Control group: no cognitive training
2. Experimental Group 1: Cognitive Training program 10 days prior to surgery.
3. Experimental Group 2: Cognitive Training program 10 days prior to surgery continuing for over a inestigatorsek after surgery.

The evaluation of the cognitive function will be carried out following the same protocol for all the three groups and will take place at different times of the perioperative period, initially on the preanesthesia visit to set a baseline, and later on the postoperative period at 3 days, 1 month and 3 month post-surgery.

Study population:

Men and women, ASA I-III, betinestigatorsen 55-70 years of age who are visited in the pre-anesthesia clinic, and scheduled for elective, noncardiac surgery, understand the purpose of the study, sign informed consent and meet the selection criteria.

Variables:

Independent: Cognitive training, through the computer application "Sincrolab". Dependent: Development of PCD, measured through the application of a neuropsychological test battery that test the cognitive domain of memory and executive functions.

The implementation of an effective program for screening, prevention and treatment of the PCD, can have a direct impact on patient safety, improve outcomes of surgical interventions and help in maintaining quality of life and active role in society of our older patients.

With the aging of the population, PCD is a problem that will become increasingly important to measure, and inestigators can imagine a multidisciplinary approach to be necessary since a patient disabled by PCD is a health problem with important economic and social connotations. Therefore, the preservation of the brain's functional and cognitive capacities deserves all of our attention and interest.

ELIGIBILITY:
Inclusion Criteria:

* >55y <70y
* Patients ASA I, II, II
* Medium or high surgical complexity

Exclusion Criteria:

* <55y
* previous surgery less than 6 month ago
* psychiatric disease
* Neurological disease
* Brain tumors
* expected survival less than 3 month
* emergencies

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Measure the effectiveness of a cognitive training program on the post op cognitive dysfunction | 3 months
  Impact of a training program on the cognitive dysfunction measured with: Mini-cog test for. Scale: 0-5, normal values > 3; measurements at 3 days, 1 month and 3 month after surgery

SECONDARY OUTCOMES:
Impact of a training program on the memory alterations | 3month
  Impact of a training program on the memory alterations measured with T@M test. Scale: 0-50. normal values > 35 and < 5 minutes execution test time.; measurements at 3 days, 1 month and 3 month after surgery
Impact of a training program on the alteration of the daily memory | 3 month
  Impact of a training program on the alteration of the daily memory measured with test: MFE Test for evaluation of the daily memory. Scale 0-84. normal values: Variations < 20%; measurements at 3 days, 1 month and 3 month after surgery
Impact of a training program on the alterations of anxiety and depression | 3 month
  Impact of a training program on the alterations of anxiety and depression measured with Goldberg Test. Anxiety scale: 0-9, normal values < 5, Depression scale: 0-9, normal values <3; measurements at 3 days, 1 month and 3 month after surgery
Measure the development of PCD in the different patient groups in relation of age | 3 month
  Measure the development of the PCD in the different patient groups in relation of the age of the patient. Measured in the different study areas: cognitive, memory, daily memory, anxiety and depression.
Measure the development of PCD in relation of sex in the different patient groups | 3 month
  Measure the development of the PCD in the different patient groups in relation of sex of the patient. Measured in the different study areas: cognitive, memory, daily memory, anxiety and depression
Measure the development of PCD in relation of duration of surgery in the different patient groups | 3 month
  Measure the development of the PCD in the different patient groups in relation of the duration of the surgery. Measured in the different study areas: cognitive, memory, daily memory, anxiety and depression
Measure the development of PCD in relation of anesthesia technique in the diferent patient group | 3 month
  Measure the development of the PCD in the different patient groups in relation of the type of anesthesia. General intravenous anesthesia, general inhalatory anesthesia, regional anesthesia. Measured in the different study areas: cognitive, memory, daily memory, anxiety and depression
Measure the development of PCD in relation of type of post operative complications, in the different patient gruops | 3 month
  Measure the development of the PCD in the different patient groups in relation of the post-operative complications. Measured in the different study areas: cognitive, memory, daily memory, anxiety and depression
Adherence to the cognitive training program | 3 month
  Assessment of the adherence to the proposed cognitive training, determining the rate of drop-outs in the PCD

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodiera Olivé, MD.Ph., Study Director — Centro Medico Teknon
Locations (1):
- Centro Medico Teknon, Servei d'anestesiologia, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steinmetz J, Rasmussen LS. Peri-operative cognitive dysfunction and protection. Anaesthesia. 2016 Jan;71 Suppl 1:58-63. doi: 10.1111/anae.13308. PMID 26620148
- [Background] Scott JE, Mathias JL, Kneebone AC. Postoperative cognitive dysfunction after total joint arthroplasty in the elderly: a meta-analysis. J Arthroplasty. 2014 Feb;29(2):261-7.e1. doi: 10.1016/j.arth.2013.06.007. Epub 2013 Jul 23. PMID 23890520
- [Background] Fong TG, Hshieh TT, Wong B, Tommet D, Jones RN, Schmitt EM, Puelle MR, Saczynski JS, Marcantonio ER, Inouye SK. Neuropsychological profiles of an elderly cohort undergoing elective surgery and the relationship between cognitive performance and delirium. J Am Geriatr Soc. 2015 May;63(5):977-82. doi: 10.1111/jgs.13383. Epub 2015 May 4. PMID 25944109
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Kawano T, Eguchi S, Iwata H, Tamura T, Kumagai N, Yokoyama M. Impact of Preoperative Environmental Enrichment on Prevention of Development of Cognitive Impairment following Abdominal Surgery in a Rat Model. Anesthesiology. 2015 Jul;123(1):160-70. doi: 10.1097/ALN.0000000000000697. PMID 26001032
- [Background] Shu AH, Wang Q, Chen XB. Effect of different depths of anesthesia on postoperative cognitive function in laparoscopic patients: a randomized clinical trial. Curr Med Res Opin. 2015;31(10):1883-7. doi: 10.1185/03007995.2015.1075968. Epub 2015 Sep 4. PMID 26202165
- [Background] Ballard C, Jones E, Gauge N, Aarsland D, Nilsen OB, Saxby BK, Lowery D, Corbett A, Wesnes K, Katsaiti E, Arden J, Amoako D, Prophet N, Purushothaman B, Green D. Optimised anaesthesia to reduce post operative cognitive decline (POCD) in older patients undergoing elective surgery, a randomised controlled trial. PLoS One. 2012;7(6):e37410. doi: 10.1371/journal.pone.0037410. Epub 2012 Jun 15. PMID 22719840
- [Background] Saleh AJ, Tang GX, Hadi SM, Yan L, Chen MH, Duan KM, Tong J, Ouyang W. Preoperative cognitive intervention reduces cognitive dysfunction in elderly patients after gastrointestinal surgery: a randomized controlled trial. Med Sci Monit. 2015 Mar 17;21:798-805. doi: 10.12659/MSM.893359. PMID 25782136